Official Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel Dose Study to

Evaluate the Safety and Efficacy of CTP-543 In Adult Patients With Moderate

to Severe Alopecia Areata

NCT Number: NCT03137381

**Document Date:** SAP Version 2: 07 May 2019

# STATISTICAL ANALYSIS PLAN 07 May 2019

# A DOUBLE-BLIND RANDOMIZED, PLACEBO-CONTROLLED STUDY TO EVALUATE THE SAFETY AND EFFICACY OF CTP-543 IN ADULT PATIENTS WITH MODERATE TO SEVERE ALOPECIA AREATA

#### PROTOCOL NUMBER CP543.2001

#### SPONSORED BY

Concert Pharmaceuticals, Inc. 99 Hayden Avenue, Suite 500 Lexington, MA 02421 Telephone: (781) 860-0045



This document is confidential and proprietary to **Concert Pharmaceuticals, Inc.** Acceptance of this document constitutes agreement by the recipient that no unpublished information contained herein will be reproduced, published, or otherwise disclosed without the prior written approval of **Concert Pharmaceuticals, Inc.**, except that this document may be disclosed to appropriate Institutional Review Boards under the condition that they keep the information confidential.

#### DOCUMENT VERSION CONTROL

Version: 2.0 

| Version Number | Date | Comments/Changes |
|----------------|-------------------|------------------|
| 0.1 | 11 September 2017 | DRAFT 1 |
| 0.2 | 20 October 2017 | DRAFT 2 |
| 0.3 | 20 February 2018 | DRAFT 3 |
| 0.4 | 10 May 2018 | DRAFT 4 |
| 1.0 | 04 June 2018 | VERSION 1.0 |
| 2.0 | 07 May 2019 | VERSION 2.0 |


#### **APPROVALS**




# TABLE OF CONTENTS

| LIS | T OF ABBREVIATIONS | 6 |
|---|---|---|
| LIS | T OF IN-TEXT TABLES | 8 |
| 1. | PURPOSE OF THE STATISTICAL ANALYSIS PLAN | 9 |
| 2. | PROTOCOL SUMMARY | . 10 |
| | 2.1 Study Objectives | . 10 |
| | 2.1.1 Primary Objective | |
| | 2.1.2 Exploratory Objectives | . 10 |
| | 2.2 Study Design | . 10 |
| | 2.3 Study Population | . 12 |
| | 2.4 Treatment Regimens | . 12 |
| | 2.5 Treatment Group Assignments or Randomization | . 12 |
| | 2.6 Sample Size Determination | |
| 3. | GENERAL ANALYSIS AND REPORTING CONVENTIONS | . 14 |
| <b>4</b> . | ANALYSIS POPULATIONS | . 16 |
| | 4.1 Efficacy Population | |
| | 4.2 Pharmacokinetic Population | |
| | 4.3 Safety Population | |
| | 4.4 Per Protocol Population | . 16 |
| <b>5</b> . | STUDY PATIENTS | . 17 |
| | 5.1 Disposition of Patients | . 17 |
| | 5.2 Protocol Deviations. | . 17 |
| <b>6</b> . | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | . 18 |
| | 6.1 Prior and Concomitant Medications | . 19 |
| <b>7.</b> | MEASUREMENTS OF TREATMENT COMPLIANCE | . 20 |
| 8. | EFFICACY EVALUATION | . 21 |
| | 8.1 Primary Efficacy Endpoint | . 21 |
| | 8.1.1 Severity of Alopecia Tool (SALT) | |
| | 8.2 Exploratory Efficacy Endpoints | |
| | 8.2.1 Visual Analog Scale (VAS) | |
| | Clinician VAS of Severity (VAS-S) | . 22 |
| | Patient VAS of Severity (VAS-S) | . 22 |
| | 8.2.2 Clinical Global Impression of Improvement (CGI-I) | . 23 |
| | 8.2.3 Patient Global Impression of Improvement (PGI-I) | . 23 |
| | 8.2.4 Patient Reported Outcomes: Alopecia Areata Symptom Impact Scal | |
| | (AASIS) and Exploratory Questions 8.3 Overview of Efficacy Analysis Issues | |
| | 8.3.1 Handling of Dropouts or Missing Data | |
| | 8.3.2 Multicenter Studies | |
| | 8.3.3 Assessment Visit Windows | |
| | 8.4 Analysis Methods | |
| | 8.4.1 Primary Efficacy Analysis | . 26 |
| | 8.4.2 Exploratory Efficacy Analyses | |
| | 8.5 Examination of Subgroups | |

| 9. | SAFETY EVALUATION | 29 |
|---|---|---|
| | 9.1 Overview of Safety Analysis Methods | 29 |
| | 9.2 Adverse Events | 29 |
| | 9.3 Clinical Laboratory Evaluation | 31 |
| | 9.4 Vital Signs, Physical Findings, and Other Observations Related to Safety | |
| | 9.4.1 Vital Signs | |
| | 9.4.2 ECG | 32 |
| | 9.4.3 Physical Examinations | |
| 10. | PHARMACOKINETIC EVALUATION | 33 |
| | 10.1 Pharmacokinetic and Pharmacodynamic Methods | 33 |
| 11. | INTERIM ANALYSES AND DATA MONITORING | 34 |
| <b>12</b> . | CHANGES TO THE ANALYSES PLANNED IN THE PROTOCOL | 35 |
| 13. | REFERENCES | 36 |
| 14. | LIST OF PLANNED TABLES | 37 |
| 15. | LIST OF PLANNED FIGURES | 44 |
| 16. | LIST OF PLANNED DATA LISTINGS | 45 |
| <b>17</b> . | APPENDICES | 47 |
| | 17.1 Study Flow Chart | 47 |
| | 17.2 Schedule of Events | |
| 18. | ATTACHMENTS | 50 |

# **LIST OF ABBREVIATIONS**

| Abbreviation or<br>Specialist Term | Explanation |
|---|---|
| AASIS | Alopecia Areata Symptom Impact Scale |
| AE | Adverse event |
| ANCOVA | Analysis of Covariance |
| ATC | Anatomical-Therapeutic-Chemical |
| BID | Twice daily dosing |
| CGI-I | Clinical Global Impression of Improvement |
| CI | Confidence interval |
| СМН | Cochran-Mantel-Haenszel Test |
| CSR | Clinical study report |
| CTCAE | Common terminology criteria for adverse events |
| DMC | Data monitoring committee |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| HDL | High-density lipoprotein |
| ICH | International Conference on Harmonisation |
| LDL | Low-density lipoprotein |
| LOCF | Last Observation Carried Forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMRM | Mixed-effects Model of Repeated Measures |
| PD | Pharmacodynamic |
| PGI-I | Patient Global Impression of Improvement |
| PK | Pharmacokinetic |
| QT | QT interval |
| QTcF | QT interval corrected for heart rate (Fridericia's method) |
| SAE | Serious Adverse Event |
| SALT | Severity of Alopecia Tool |
| SAP | Statistical Analysis Plan |
| SD | Standard deviation |
| SOC | System organ class |


| TEAE | Treatment-emergent adverse events |
|----------|-----------------------------------|
| VAS-S | Visual Analog Scale of Severity |
| WHO | World Health Organization |
| $\chi^2$ | Chi-squared test |


| ı | IST | OF | IN- | <b>TEXT</b> | TAF | 31 FS |
|---|-----|--------|-----|-------------|-----|-------|
| - | | $\sim$ | _ | | | |

| Table 8-1 | Efficacy ' | Variables | and Analysis | Methods | <br>25 |
|-----------|------------|-----------|---------------|-----------|--------|
| | Lilloacy | v anabics | and / marvois | INICHIOGS | <br> |


#### 1. PURPOSE OF THE STATISTICAL ANALYSIS PLAN

This statistical analysis plan (SAP) contains detailed information to aid in the implementation of the statistical analyses and reporting of the study data for use in the clinical study report (CSR) for study CP543.2001. This SAP is being written with due consideration of the recommendations outlined in the most recent International Conference on Harmonisation (ICH) E9 Guideline, entitled Guidance for Industry: Statistical Principles for Clinical Trials, and the most recent ICH E3 Guideline, entitled Guidance for Industry: Structure and Content of Clinical Study Reports.

This SAP describes the data sets that will be used for analysis, as well as patient characteristics, efficacy, safety, pharmacokinetic (PK), pharmacodynamic (PD), and clinician-reported and patient-reported perception of disease severity and improvement parameters. The details of the specific statistical methods stated in the protocol will be provided and any changes from the protocol-specified analyses will be documented in the SAP prior to database lock. Pharmacokinetic analyses are outside the scope of this document and will be performed and reported separately. If additional analyses are required to supplement the planned analyses described in this SAP after the database lock, they may be completed and will be described in the CSR. Table, figure, and listing specifications are provided as an attachment in a separate document. The CP543.2001 protocol amendment 2.0 was finalized on 05 July 2017. The purpose of this amendment was to revise for a new sequential cohort study design, where a parallel active dose comparison would no longer be conducted. Amendment 3.0, dated 25 September 2017, further clarifies this revised approach. Amendment 4.0, dated 17 August 2018, included an additional Cohort of subjects to assess a 12 mg BID dose of CTP-543 compared to placebo. The sample size calculations were updated to reflect the additional patients enrolled. Amendment 5.0, dated 21 January 2019, included language for allowing eligible patients who completed dosing for 24 weeks to enter an open-label extension study of CTP-543. This SAP is based on the latest protocol amendment.


#### 2. PROTOCOL SUMMARY

## 2.1 Study Objectives

The overall objectives of the study are to assess the safety and efficacy of a 24-week regimen of administration of CTP-543 in adult patients with chronic, moderate to severe alopecia areata.

# 2.1.1 Primary Objective

- To assess the effect of CTP-543 on treating hair loss as measured by the Severity of Alopecia Tool (SALT);
- To assess the safety of administration of CTP-543 in adult patients with chronic, moderate to severe alopecia areata.

# 2.1.2 Exploratory Objectives

- To assess the change in alopecia areata severity as measured by the clinician Visual Analog Scale of Severity (VAS-S) from baseline;
- To assess the Clinical Global Impression of Improvement (CGI-I);
- To assess the change in alopecia areata severity as measured by the patient VAS-S from baseline;
- To assess the Patient Global Impression of Improvement (PGI-I);
- To assess the change in patient reported outcomes as measured by the Alopecia Areata Symptom Impact Scale (AASIS) and exploratory questions from baseline.

# 2.2 Study Design

This is a double-blind, randomized, placebo-controlled multicenter study to evaluate the safety and efficacy of CTP-543 in adult patients with chronic, moderate to severe alopecia areata. Patients will be between 18 and 65 years of age and experiencing an episode of alopecia areata lasting at least 6 months and not exceeding 10 years, with at least 50% hair loss as measured by the SALT at Screening and Baseline, and are not concurrently being treated for alopecia areata or with other treatments that might affect hair regrowth or immune response. Approximately 50% of alopecia areata patients with alopecia totalis or universalis, and approximately 10% with only alopecia ophiasis will be enrolled.

The study consists of up to 3 cohorts initiated sequentially in ascending dose order. An independent data monitoring committee (DMC) will determine if there are adequate safety data to support each subsequent higher dose cohort. Patients will not dose escalate within a cohort and may only participate in one cohort.


The Screening Period may last up to 28 days prior to randomization and initiation of study drug. The Treatment Period is the initial 24-week, double-blind, placebo-controlled period to define efficacy and safety of CTP-543 compared to placebo. The Post-Treatment Safety Follow-up Period is the final 4 weeks of each cohort to assess safety following treatment completion. Patients enrolled in Cohort 3 (12 mg BID) will have the option to continue receiving treatment in an open-label extension study following the treatment period. If patients do not wish to continue into the open-label extension study, they will complete treatment at Week 24 and return in 4 weeks for the Post-Treatment Safety Follow-up to assess safety following treatment completion.

The DMC will perform regular safety assessments for each cohort based on review of collective safety data. After the last patient has completed the Week 12 Visit within a cohort, the DMC will convene to review accumulated safety data to assess if initiation of the subsequent cohort is supported. The DMC may advise treatment arm cessation due to intolerability at any time.

Patients will provide appropriately obtained informed consent prior to completing any screening procedures. Patients meeting screening criteria will be eligible to continue to the Day 1 visit for review of eligibility and baseline assessments, including SALT, physical examination, clinical laboratory assessments, vital signs, and electrocardiogram (ECG). For each cohort, patients meeting all inclusion criteria and none of the exclusion criteria will be randomized to CTP-543 treatment or placebo. The first 2 cohorts will be randomized in a 2:1 ratio (active:placebo) and the third cohort will be randomized in a 5:1 ratio (active:placebo) in order to provide a similar number of patients across each CTP-543 dose and overall placebo (pooled) group. Randomization will be stratified by classification of alopecia areata subtype into one of the following three categories: 1) alopecia areata, 2) alopecia totalis or alopecia universalis, or 3) alopecia ophiasis.

The double-blind, placebo-controlled Treatment Period for each cohort will last 24 weeks. Assessment of treatment response with SALT for efficacy will occur at 4, 8, 12, 16, 20 and 24 weeks. The final efficacy analysis will be conducted when all patients in the 12 mg cohort have completed Week 24.

For Cohorts 1 and 2, patients will stop taking study medication upon completion of treatment at Week 24 and enter a 4-week Post-Treatment Safety Follow-Up Period. Patients will be assessed for safety through Week 28. For Cohort 3, patients will either complete treatment at Week 24 and have a Safety Follow-up visit at Week 28 prior to exiting the study, or if eligible, may enroll into an Open-label Extension study of CTP-543 at their Week 24 visit.

Patients enrolled into each cohort will take the first dose of study drug in the clinic on Day 1 and will be instructed to take study drug every 12 hours for the duration of the Treatment Period. Patients will dose study drug in the clinic on all Study Visit Days after clinical laboratory blood draws are completed. Blood samples for pharmacokinetic and pharmacodynamic assessment will be taken periodically. Scheduled assessment of patient and clinician perception of disease


severity and improvement will also occur. Patient safety will be monitored throughout the trial and supported by regular review by the DMC.

Hematology parameters will be monitored closely for the duration of the study. For each cohort, hematology will be conducted every 2 weeks during the first 8 weeks of the Treatment Period, followed by an assessment every 4 weeks thereafter through completion of the study. Lipid levels will be assessed every 12 weeks throughout the Treatment Period and at the Post-Treatment Safety Follow-Up Visit, if applicable. Significant cytopenias or other hematologic abnormalities will be managed by dose interruption and signs and symptoms of infection will be treated promptly. Patients who experience intolerable symptoms during treatment may discontinue the study at the discretion of the Investigator. Patients may withdraw consent at any time.

# 2.3 Study Population

The study population will consist of male and female patients of any ethnicity between 18 and 65 years of age, inclusive, with diagnosis of alopecia areata with a current episode lasting at least 6 months and not exceeding 10 years at the time of Screening. Total disease duration greater than 10 years is permitted. Patients must also exhibit at least 50% scalp hair loss, as defined by a  $SALT \ge 50$ , at Screening and Baseline.

A full list of the inclusion and exclusion criteria can be found in Sections 8.1 and 8.2 in the CP543.2001 Protocol.

# 2.4 Treatment Regimens

CTP-543 will be dosed orally as tablets at doses 4 mg, 8 mg, 12 mg, or matching placebo, every 12 hours during the Treatment Period. Doses will be allocated to each cohort as follows:

- Cohort 1: 4 mg (2:1 CTP-543 4 mg : placebo)
- Cohort 2: 8 mg (2:1 CTP-543 8 mg : placebo)
- Cohort 3: 12 mg (5:1 CTP-543 12 mg : placebo)

#### 2.5 Treatment Group Assignments or Randomization

Patients meeting all inclusion criteria and none of the exclusion criteria will be randomized to CTP-543 treatment or placebo. The first 2 cohorts will be randomized in a 2:1 ratio (active:placebo) and the third cohort will be randomized in a 5:1 ratio (active:placebo) in order to provide a similar number of patients across each CTP-543 dose and the overall placebo (pooled) group. Randomization will be stratified by classification of alopecia areata subtype into one of the following three categories: 1) alopecia areata, 2) alopecia totalis or alopecia universalis, or 3)


alopecia ophiasis. Approximately 50% of alopecia areata patients with alopecia totalis or universalis, and approximately 10% with only alopecia ophiasis will be enrolled.

## 2.6 Sample Size Determination

There are very few studies in the literature to provide reliable estimates of active treatment or placebo response rates using SALT, or the estimate of variances around these measures, in patients with alopecia areata. Power calculations assume a 2-sided chi-squared test and significance level of 0.05 and are based on an active treatment response rate of 45% and a placebo response rate of 10%.

Although patients will be randomized in an unbalanced ratio of active drug to placebo within each cohort, the placebo patients from the 3 cohorts will be combined for statistical comparisons to each active treatment group. The first 2 cohorts will be randomized in a 2:1 ratio (active:placebo) and the third cohort will be randomized in a 5:1 ratio (active:placebo). Based on estimated completion rates, this randomization scheme is expected to provide a similar number of patients in each CTP-543 dose group and the pooled placebo group. Thus, power calculations for the comparison to placebo are based on a 1:1 treatment ratio of each CTP-543 dose group to placebo. Power calculations assume a 2-sided test and significance level of 0.05 and are based on an active treatment response rate of 45% and a placebo response rate of 10%. Based on estimated completion rates as of Amendment 4, this randomization scheme is expected to provide a similar number of patients in the 12 mg group and the pooled placebo group.

A sample size of 28 patients in the 12 mg group and 28 patients in the pooled placebo group will provide >80% power for the chi-squared test when comparing each dose group to the combined placebo group (28 active, 28 placebo). Approximately 150 patients will be randomized in order to provide 120 patients who complete treatment.


#### 3. GENERAL ANALYSIS AND REPORTING CONVENTIONS

The following is a list of general analysis and reporting conventions to be applied to this study, unless otherwise specified.

All data displays (tables, listings, and figures) will have a header showing the sponsor company name, protocol number, page number, and display status (i.e. "DRAFT" or "FINAL"), as well as a footer indicating path, file name, and run date/time. Summary tables and data listings will be summarized by treatment and overall, as appropriate. All data collected per-protocol and all derived variables will be listed

Categorical variables will be summarized using counts (n) and percentages (%) and will be presented in the form "n (xx.x)." If a count is 0, 0% will be shown for the percentage. If a percentage is 100%, 100% will be shown with no decimal place. To ensure completeness, summaries for categorical variables will include all categories, even if no patients had a response in a particular category. Unless otherwise specified, the denominator for each percentage will be based on the number of patients in the population being summarized (header n). If missing values are present, counts will be shown but will not be included in percentage calculations.

Continuous variables will be summarized using mean, standard deviation (SD), minimum, maximum, median, and number of patients. The mean and median will be reported to an additional level of precision than the original observations, and the SD will be reported to two additional levels of precision than the original observations. The minimum and maximum will be the same precision as the original data. In general, any calculated values, such as those due to unit conversion, will be rounded to the same number of decimal places as the original data.

All statistical tests will be 2-sided with a significance value of 0.05. Testing will be performed only for the Treatment Period. Estimates and confidence intervals will be reported to 1 more decimal than the original data. P-values will be reported to 3 decimal places.

Summary tables and data listings:

- No preliminary rounding will be performed; rounding will only occur after analysis.
- Data from patients excluded from an analysis population will be presented in the data listings but will not be included in the calculation of summary statistics, where applicable.
- Data from each patient will be separated by a blank line. Within a data listing, if a
  descriptive item appears line after line (e.g., repetition of a patient number, date, visit,
  etc.), only the first occurrence will be displayed (e.g., in Listing of Vital Signs, patient
  number, date and visit will only be displayed on first row when presenting all parameters


collected at same visit). Repetition of actual results or outcomes (e.g., Adverse Events (AEs), lab results, vital sign values, etc.) will not be collapsed.

- Data listings will be sorted by cohort within treatment, patient, and week and/or time of assessment, as applicable.
- Placebo groups will be separated by cohort within data listings and pooled within summary tables.
- When change from baseline is calculated, baseline is the last observation obtained prior to dosing of the study drug.

Mock tables and data listings will be provided as attachments to this analysis plan. Minor changes to the mocks after formal SAP approval will not necessitate re-approval unless changes to the text of the SAP are required.

All statistical deliverables will be produced, validated, and reviewed for accuracy/consistency in accordance with standard operating procedures and the processes described in the statistical validation plan.

SAS® (SAS Institute, Cary, North Carolina) statistical software, version 9.4 or later, will be used for all analyses. Adverse Events and Medical History will be coded in Medical Dictionary for Regulatory Activities (MedDRA) Version 19.1. Concomitant medications will be coded in World Health Organization (WHO) Drug Version E (2016.01) and Anatomical-Therapeutic-Chemical (ATC) classification and preferred term.


#### 4. ANALYSIS POPULATIONS

Analysis populations will be summarized and listed for each patient, by treatment and cohort.

# 4.1 Efficacy Population

The Efficacy Population will include all patients who receive study drug and have at least 1 post-treatment SALT assessment during the Treatment Period. Patients in the Efficacy Population will be analyzed according to their randomized treatment group.

#### 4.2 Pharmacokinetic Population

The Pharmacokinetic Population will include all patients who receive study drug and have at least 1 pharmacokinetic sample taken during the Treatment Period. Patients who receive placebo will be excluded from the Pharmacokinetic Population.

# 4.3 Safety Population

The Safety Population will include all patients who receive study drug during the Treatment Period. Patients in the Safety Population will be analyzed according to the actual treatment received during the study.

## 4.4 Per Protocol Population

The Per Protocol Population will include all patients in the Efficacy Population who were dosed according to protocol, have a week 24 SALT score, and have no major protocol deviations. The procedure for defining major protocol deviations is described in Section 5.2.


#### 5. STUDY PATIENTS

# 5.1 Disposition of Patients

Disposition will be summarized by randomized treatment group for all patients screened in the study. The following disposition information will be summarized (percentages based on the number randomized, with the exception of the reasons for discontinuation):

- The number of patients screened.
- The number of patients randomized.
- The number and percentage of patients treated within the Efficacy, Pharmacokinetic, Safety, and Per Protocol Populations.
- The number and percentage of patients who completed the study (defined as completing all study visits) and who completed 24 weeks of treatment.
- The number and percentage of patients who prematurely discontinued, and the frequency and percentage of each discontinuation reason. The denominator for the percentage of each discontinuation reason will be the number of patients who discontinued.

Disposition and patient visits will also be presented for each patient in patient data listings. Patient data listings will list date of informed consent, date of first/last treatment, date of end of study/early termination, and reasons for discontinuation. Additionally, screen failures post and prior to Amendment 2 will be presented in separate listings. A Kaplan Meier curve of time to last dose will also be presented.

#### 5.2 Protocol Deviations

Protocol deviations will be collected at both the site and patient level on the Electronic case report form (eCRF). A blinded data review will be conducted before database lock by the sponsor to classify protocol deviations as minor or major. Deviations that may alter or confound interpretation of the study results will be classified as major deviations. Protocol deviations will be summarized by deviation classification and category for all randomized patients and listed by patient in a data listing. Protocol deviations that are identified as major will be used to exclude patients from the Per Protocol population.


#### 6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Demographic characteristics (i.e., sex, ethnic origin, race, date of birth, and calculated body mass index) will be collected at the Screening Visit, between Day -28 and -1, and detailed on the eCRF.

The patient's alopecia areata will be classified by the Investigator into one of three categories defined for this study:

- 1) Alopecia areata: patchy type hair loss,
- 2) Alopecia totalis or universalis: complete hair loss on the scalp with or without body hair loss,
- 3) Alopecia ophiasis: band-like hair loss limited to the periphery of the scalp along the back of the hair line in the occipital region and possibly extending over each ear in temporal regions.

The alopecia totalis and alopecia universalis category will be separated into each individual subtype for summaries. Alopecia areata category at baseline defined as the current episode and alopecia areata category at disease onset will be summarized. In addition, baseline SALT score will be presented as a baseline characteristic. The duration of the current episode in months and the duration of disease in months will also be summarized.

Duration of current episode will be calculated as: (date of randomization – date of current episode onset + 1) / 30.4375.

Duration of disease at onset will be calculated as: (date of randomization – date of disease onset + 1) / 30.4375.

All demographics and baseline characteristics will be summarized for all randomized patients with descriptive statistics and listed within a by-patient data listing.

Thorough medical history, including current medications, nail and facial hair involvement, comorbidities, as well as history of vaccination against herpes zoster collected at the Screening and Randomization Visits, will be summarized and listed.

Medical history will be summarized by frequencies of System Organ Class (SOC) and preferred term and will be coded using MedDRA Version 19.1. All medical history for each patient will be included in a data listing.


#### 6.1 Prior and Concomitant Medications

Prior and concomitant medications will be summarized by WHO Drug ATC classification level 2 and preferred term and listed within a by-patient data listing.

Medications are classified as prior if started and stopped prior to the first dose date of study drug or as concomitant if used on or after the first dose date of study drug. Concomitant medications will be recorded from Screening through the Follow-Up Visit at Week 28.

Partial and completely missing dates will be imputed for the purposes of classifying concomitant medications as follows:

- Partial dates will be imputed following the same algorithm as in 9.2 for Treatmentemergent adverse events (TEAEs).
- For an entirely missing start date (i.e. day, month, and year are missing), the start date
  will be set to the date of administration of study drug unless the stop date is prior to the
  date of administration of study drug, in which case the start date will be set to the stop
  date.

For an entirely missing stop date (i.e. day, month, and year are missing), the medication will be treated as ongoing.


#### 7. MEASUREMENTS OF TREATMENT COMPLIANCE

Patients will strive for 100% compliance with the daily dosing schedule. Treatment compliance will be summarized as time on treatment as well as percent of planned dose received for each treatment group. Time on treatment will be defined as date of last dose in the treatment period minus the date of first dose in the treatment period + 1. Percent of planned dose received will be calculated for the entire treatment period as follows:

$$100*\frac{Tablets\ Dispensed-Tablets\ Returned}{Tablets\ Expected}$$

Tablets Expected is defined as the time on treatment multiplied by the expected number of active dose pills taken daily (x2 for the 4 mg cohort, x2 for the 8 mg cohort, and x 2 for the 12 mg cohort). Dose interruptions will be ignored in this calculation. Patient compliance and dosing exceptions will be listed in by-patient data listings.


#### 8. EFFICACY EVALUATION

## 8.1 Primary Efficacy Endpoint

The primary efficacy endpoint will be the proportion of responders, defined as patients achieving at least a 50% relative reduction in SALT score, from baseline at Week 24.

#### 8.1.1 Severity of Alopecia Tool (SALT)

The SALT is a measure of hair absence that quantifies the amount of scalp surface without hair in a pre-specified quadrant of the scalp (right side, top, left side, back), that is further summed after applying a quadrant-specific multiplier indicative of scalp surface area contribution, to provide an overall score of total hair loss. Total SALT score is computed as [(left quadrant raw score x 0.18) + (right quadrant raw score x 0.18) + (top quadrant raw score x 0.40) + (back quadrant raw score x 0.24)]. The SALT assessment will occur via live examination of the patient during clinic visits.

As the SALT score is by nature a measurement of total surface without hair, it is important to note that in the context of this SAP, endpoints will follow these definitions:

- Absolute change = difference in SALT measurements (follow-up SALT score minus baseline SALT score)
- Relative change = percent change of the follow-up SALT score, where baseline SALT score is the denominator (i.e. absolute change divided by the baseline score, multiplied by 100)

# 8.2 Exploratory Efficacy Endpoints

Exploratory efficacy endpoints include:

- The proportion of responders at Weeks 4, 8, 12, 16 and 20;
- Proportion of responders who have at least 75%, 90% and 100% relative reduction in SALT score from baseline at Weeks 4, 8, 12, 16, 20, and 24;
- Absolute change in SALT scores from baseline at Weeks 4, 8, 12, 16, 20, and 24 in the Blinded Treatment Period;
- Relative change in SALT scores from baseline at Weeks 4, 8, 12, 16, 20, and 24 in the Blinded Treatment Period:
- Absolute SALT scores at Weeks 4, 8, 12, 16, 20, and 24 in the Blinded Treatment Period;
- Proportion of patients achieving an absolute SALT score of  $\leq$ 10,  $\leq$ 20, and  $\leq$ 25 at Weeks 4, 8, 12, 16, 20 and 24;
- Percent change in alopecia areata severity from baseline as measured by the clinician VAS-S at Weeks 12 and 24;


- Changes in alopecia areata from baseline as measured by the clinician rated 7-point Likert scale CGI-I at Weeks 12 and 24;
- Proportion of subjects worsening in alopecia areata from baseline to Weeks 12 and 24 as measured by responses of "Very Much Worse" or "Much Worse" on the clinician rated CGI-I;
- Proportion of subjects improving from baseline to Weeks 12 and 24 as measured by responses of "Very Much Improved" or "Much Improved" on the clinician rated CGI-I;
- Percent change in alopecia areata severity from baseline as measured by the patient VAS-S at Weeks 12 and 24;
- Changes in alopecia areata from baseline as measured by the patient rated 7-point Likert scale PGI-I at Weeks 12 and 24;
- Proportion of subjects worsening in alopecia areata from baseline to Weeks 12 and 24 as measured by responses of "Very Much Worse" or "Much Worse" on the patient rated PGI-I;
- Proportion of subjects improving from baseline to Weeks 12 and 24 as measured by responses of "Very Much Improved" or "Much Improved" on the patient rated PGI-I;
- Patient-reported outcomes: Changes in symptoms from baseline as measured by AASIS and exploratory questions at Week 24.

# 8.2.1 Visual Analog Scale (VAS)

The VAS is a scale initially developed for pain that has been used in a variety of clinical settings where the endpoint of interest is based on patient perception. The VAS is a distinct 100 millimeter line anchored on the left end at full degree of impairment and on the right end at no degree of impairment, where indication of the degree of impairment perceived at the time of assessment is captured by marking the appropriate position on the line between the anchor points. The measured distance of the mark from the left anchor will be recorded in millimeters. Since the VAS was measured right to left in terms on increasing impairment, the VAS analysis value will be calculated by taking 100 minus the collected value.

#### Clinician VAS of Severity (VAS-S)

The Investigator will complete a VAS-S regarding the severity of the patient's alopecia areata at the time of completion as indicated in the Schedule of Events. The left and right anchor points for the clinician VAS-S are "Extremely Apparent" and "Not At All Apparent", respectively.

#### Patient VAS of Severity (VAS-S)

Patients will rate perception of his/her alopecia areata severity on the patient VAS-S. The left and right anchor points for the patient's alopecia areata VAS-S are "Extremely Apparent" and


"Not At All Apparent", respectively. The patient VAS-S will measure the patient's perception of his/her alopecia areata at the time of completion.

## 8.2.2 Clinical Global Impression of Improvement (CGI-I)

Compared to the patient's alopecia areata prior to treatment at baseline, the patient's current state of alopecia areata will be assessed according to the Investigator's perceived change. The Investigator may select one of seven numeric choices from 1 to 7, with 1 representing "Very Much Improved" to 7 representing "Very Much Worse".

#### 8.2.3 Patient Global Impression of Improvement (PGI-I)

Compared to the patient's alopecia areata prior to treatment at baseline, the patient's current state of alopecia areata will be assessed according to his/her perceived change. The patient may select one of seven numeric choices from 1 to 7, with 1 representing "Very Much Improved" to 7 representing "Very Much Worse".

# 8.2.4 Patient Reported Outcomes: Alopecia Areata Symptom Impact Scale (AASIS) and Exploratory Questions

The AASIS is a questionnaire designed to measure the quality of life, symptoms, and their impact for patients with alopecia areata [Mendoza 2013]. Three dimensions related to alopecia areata are assessed: impact of alopecia areata, hair loss, and physical skin symptoms. All responses will be summed to produce the AASIS score.

In addition to the AASIS, exploratory questions will be used to attempt to define clinically meaningful outcomes for patients with alopecia areata.

## 8.3 Overview of Efficacy Analysis Issues

# 8.3.1 Handling of Dropouts or Missing Data

The Last Observation Carried Forward (LOCF) approach will be implemented for missing SALT score data, e.g., if the SALT score in the Week 16 visit window is missing, the next and closest available on-treatment SALT score measurement before the Week 16 visit window will be used for all remaining SALT assessments: Week 16, Week 20 and Week 24. Missing baseline values will not be carried forward. If a SALT assessment is missing between two non-missing SALT


assessments visits, the SALT score at that visit will be interpolated using the mean of the closest pre- and post-assessments.

If the number of discontinuations due to adverse events is substantial, other methods will be explored.

#### 8.3.2 Multicenter Studies

Patients will be enrolled at up to 15 sites. To reduce variability, one rater should perform each clinician dependent assessment (SALT, VAS-S, and CGI-I) for the patient for the duration of the study. All investigators using the SALT will be trained prior to use.

#### 8.3.3 Assessment Visit Windows

The visit schedule for all study assessments is provided in appendix 17.2. Patients will be considered completed for efficacy analyses after Week 24 (Visit 10). For Cohorts 1 and 2, patients will stop taking study medication upon completion of treatment at Week 24 and enter a 4-week Post-Treatment Safety Follow-Up Period. For Cohort 3, patients will either complete treatment at Week 24 and have a Safety Follow-up visit at Week 28 prior to exiting the study, or if eligible, may enroll into an Open-label Extension study of CTP-543 at their Week 24 visit.

For scheduled visits, there will be no reassignment of the analysis visit based on date, and all data will appear in summary tables based on the nominal timepoint.

Unscheduled and repeat safety visits will be assigned to the closest prior planned visit. If the closest planned visit is already documented, the unscheduled or repeat visit will only be listed and will not be summarized.

# 8.4 Analysis Methods

All statistical tests will be 2-sided with a significance value of 0.05. Testing will be based on the Efficacy population and performed only for the Treatment Period. An analysis of the primary efficacy endpoint and exploratory SALT endpoints will also be performed for the Per Protocol population. The final efficacy analysis will be conducted when all patients in the 12 mg cohort have completed Week 24. The placebo groups from all 3 cohorts will be pooled and compared to each active dose (4 mg, 8 mg, and 12 mg) individually. Active doses, 4 mg, 8 mg, and 12 mg, will also be compared. There will be no adjustment for multiple treatment group comparisons in this dose-ranging Phase 2 study.

Table 8-1 gives an overview of the analysis methods that will be used for each of the efficacy variables.


Table 8-1 Efficacy Variables and Analysis Methods

| Efficacy Variables | <b>Collection Times</b> | Method |
|---|---|---|
| Primary | | |
| Responder Analysis | Baseline, Week 24 | $\chi^2$ Test |
| SALT (50% relative reduction) | | |
| Exploratory | | |
| Responder Analysis<br>SALT (50% relative reduction) | Baseline, Week 4, 8, 12, 16, 20 | $\chi^2$ Test |
| Responder Analysis<br>SALT (75%, 90%, and 100%<br>relative reduction) | Baseline, Week 4, 8, 12, 16, 20, 24 | $\chi^2$ Test |
| SALT ( $\leq$ 10, $\leq$ 20, $\leq$ 25 absolute score) | Baseline, Week 4, 8, 12, 16, 20, 24 | $\chi^2$ Test |
| SALT (absolute change) | Baseline, Week 4, 8, 12, 16, 20, 24 | MMRM |
| SALT (relative change) | Baseline, Week 4, 8, 12, 16, 20, 24 | MMRM |
| SALT (absolute score) | Baseline, Week 4, 8, 12, 16, 20, 24 | MMRM |
| Clinician VAS-S (percent change) | Baseline, Week 12, 24 | ANCOVA |
| Patient VAS-S (percent change) | Baseline, Week 12, 24 | ANCOVA |
| CGI-I | Week 12, 24 | $\chi^2$ Test |
| CGI-I Responder ("Very<br>Much/Much Improved" and<br>"Much/Very Much Worse") | Week 12, 24 | $\chi^2$ Test |
| PGI-I | Week 12, 24 | $\chi^2$ Test |
| PGI-I Responder ("Very<br>Much/Much Improved" and<br>"Much/Very Much Worse") | Week 12, 24 | $\chi^2$ Test |
| AASIS | Baseline, Week 24 | Descriptive Statistics |
| Exploratory Questions | Baseline, Week 24 | Descriptive Statistics |
| Responder Analysis, Exploratory<br>Questions, Satisfied v.<br>Unsatisfied | Baseline, Week 24 | $\chi^2$ Test |

 $<sup>\</sup>chi^2$  = Chi-Squared Test; ANCOVA = analysis of covariance; CMH = Cochran-Mantel-Haenszel; MMRM = mixed-effect model for repeated measures


# 8.4.1 Primary Efficacy Analysis

The aim of this study is to demonstrate that in terms of the primary efficacy endpoint, 50% relative reduction in SALT score at Week 24, CTP-543 is superior to the placebo. Pairwise treatment group differences will be assessed with the  $\chi^2$  test.

The active treatment will be considered effective if  $p \le 0.05$ .

Number and percentage, as well as p-values based on the  $\chi^2$  test, will be reported for the responders, defined as a patient meeting at least 50% relative reduction in SALT score at Week 24. Additionally, the number and percentage of responders will be reported by alopecia areata subtype.

Responders will be presented graphically by treatment group as a bar graph at 24 Weeks and as a line graph across time.


## 8.4.2 Exploratory Efficacy Analyses

Treatment differences for absolute score, absolute change, and relative change in SALT score from baseline to Weeks 4, 8, 12, 16, 20, and 24 will be assessed with a mixed-effect model of repeated measures (MMRM). The model will include fixed factors for treatment group, study visit, treatment by study visit interaction, and alopecia areata subtype, with baseline SALT score as a covariate. An unstructured variance-covariance matrix will be used. If convergence is not achieved, an alternative autoregressive covariance structure will be used. If the MMRM model does not converge, other covariance structures will be explored. If convergence is still not met, only descriptive statistics will be presented.

Point estimates and standard errors will be presented for each treatment group at each time point. P-values for the treatment by visit interaction will be presented at Week 24 for each active treatment compared to the placebo. A comparison of the active doses (4 mg vs. 8 mg, 4 mg vs. 12 mg, 8 mg v. 12 mg) will be presented as well. Treatments will be compared overall and by visit.

Descriptive statistics will be reported for the SALT score at each time point for each treatment group and by subtype. By-patient data listing will also be presented for patient SALT scores and collection of SALT photographs. The mean of observed value, absolute change, and relative change SALT scores along with standard errors for each treatment group will be presented using line graphs.

Responders, as defined for the primary endpoint, will be analyzed per section 8.4.1 for Weeks 4, 8, 12, 16, and 20. Additionally, the following responder groups will be analyzed per section 8.4.1 at Weeks 4, 8, 12, 16, 20, and 24: 1) patients who meet at least 75%, 90%, and 100% relative change; 2) patients who meet an absolute SALT score of  $\leq$ 10,  $\leq$ 20, or  $\leq$ 25.

The percent change in clinician and patient VAS-S from baseline will be assessed using the analysis of covariance (ANCOVA) for Week 12 and 24 with fixed factors for treatment, alopecia areata subtype, and baseline VAS-S. The least squares mean score estimates with 95% CI will be presented along with p-values for each treatment comparison at each time point. Descriptive statistics will also be reported by treatment and subtype.

A  $\chi^2$  trend test will be used to analyze CGI-I and PGI-I between treatment groups overall. Responses for PGI-I and CGI-I categorized as achieving "Very Much/Much Improved" or "Much/Very Much Worse" will also be compared between treatment groups with the  $\chi^2$  test. Descriptive statistics and by-patient data listings will also be presented for the 7 response categories for each assessment.

Mean and mean change from baseline for total AASIS score will be reported. Number and percentage of subjects in each response category of AASIS will also be summarized. Individual responses will be listed in categories of "Severity" and "Interference".


The exploratory questions will be summarized with descriptive statistics at baseline and Week 24, and will be listed in the by-patient data listings. Responses will be categorized as "Satisfied" (including responses of "Very satisfied" and "Satisfied") and "Unsatisfied" (including responses of "Unsatisfied" and "Very unsatisfied") and presented as a 2 x 2 shift table from baseline to Week 24, compared with a  $\chi^2$  Test by cohort.

# 8.5 Examination of Subgroups

Descriptive statistics will be provided by alopecia subtype.


#### 9. SAFETY EVALUATION

## 9.1 Overview of Safety Analysis Methods

Safety and tolerability of CTP-543 will be assessed by evaluating the following for the Safety Population:

- Adverse events
- Clinical laboratory results
- Vital signs
- ECG results
- Concomitant medications
- Physical examinations

All safety summaries will be descriptive with no statistical hypothesis testing and based on the Safety Population. Patients will be summarized according to the study drug received (i.e., as treated), should it differ from the randomized treatment arm. All safety endpoints will be listed in by-patient data listings.

#### 9.2 Adverse Events

Adverse events will be coded using MedDRA and summarized by system organ class and preferred term. Clinically significant deteriorations in physical examination findings will be reported and summarized as adverse events.

An adverse event reported after informed consent, but before the first dose of study drug (i.e., Day 1), will be considered a pre-treatment adverse event. Treatment-emergent adverse events will be defined as any adverse event that occurs after administration of the first dose of study drug. The number and percentage of patients who report TEAEs will be summarized by system organ class and preferred term.

Treatment emergent adverse events will also be summarized by intensity as well as relationship to study drug.

Partial dates will be imputed for the purposes of defining TEAEs as follows:

• For a missing start day where the month and year are present, the start day will be set to the first day of the month, unless 1) the first day of the month is before the date of


administration of study drug and the month and year are the same as the month and year of the date of administration of study drug, and 2) the end date is on or after the date of administration of study drug or the end date is completely missing, in which case the start day will be set to the first day of administration of study drug.

- For a missing start day and month where the year is present, the start day and month will be set to January 1<sup>st</sup>, unless 1) January 1st is before the date of administration of study drug, and 2) the end date is on or after the date of administration of study drug or the end date is completely missing, in which case the start day and month will be set to that of the first date of administration of study drug.
- For a missing end day where the month and year are present, the end day will be set to
  the last day of the month, unless the month and year are the same as the month and year
  of the last contact date for the patient, in which case the end day will be set to that of the
  patient's last contact date.
- For a missing end day and month where the year is present, the end day and month will be set to the patient's last contact date, unless the year of the patient's last contact date is greater than the end year, in which case the end day and month will be set to December 31st.

For an entirely missing stop date (i.e. day, month, and year are missing), the TEAE will be treated as ongoing.

Patients who report the same preferred term on multiple occasions will be counted once for the preferred term: under the highest severity when summarized by severity and under the closest relationship to study drug when summarized by relationship. Missing severity or relationship will not be imputed. If a patient reports multiple preferred terms for a SOC, the patient will be counted only once for that SOC.

The number and percentage of patients who experience TEAEs will be summarized by treatment group for the following:

- By SOC and preferred term
- By severity/intensity, SOC, and preferred term
- By relationship to study drug, SOC, and preferred term
- Serious adverse events (SAEs) by SOC and preferred term
- SAEs by relationship to study drug, SOC and preferred term


- AEs resulting in discontinuation of study drug by SOC and preferred term
- AEs that result in study drug dose interruption by SOC and preferred term
- AEs that meet Grade 3-4 Common terminology criteria for adverse events (CTCAE) hematology results by system organ class and preferred term
- AEs that meet Grade 3-4 CTCAE serum chemistry results by system organ class and preferred term

By-patient listings will be provided for all AEs, SAEs, and AEs related to the study drug, as well as AEs leading to study drug withdrawal or death. A by-patient listing will also be created for any pregnancies that occur. TEAEs that result in dose interruption will also be identified.

Additionally, TEAEs will be summarized by time interval: 0 to 12 weeks, and 12 to 24 weeks. For each time interval, an incidence table will summarize only TEAEs with an onset date within the interval and a prevalence table will summarize all TEAEs that have an onset date within the interval or continue into the interval. Differences between the incidence and prevalence tables can provide insight into the duration of TEAEs as well as the recurrence of TEAEs. A preferred term for an individual patient will be reported in multiple time intervals if there are multiple adverse event reports. The denominator for each time interval will be the number of patients who received at least 1 dose of study drug within the interval. These incidence and prevalence tables will be repeated for key hematology and serum chemistry AEs categorized as CTCAE Grade 3-4 results.

# 9.3 Clinical Laboratory Evaluation

Observed measurements along with change from baseline for each scheduled assessment will be summarized descriptively by treatment group and visit for each clinical laboratory parameter.

Hematology parameters for patients that meet Grade 3 or Grade 4 toxicity criteria from the CTCAE v4.0 for neutrophils, platelets, and hemoglobin will be summarized for each scheduled visit and overall for all post-baseline visits. In addition, hematology parameters of interest that meet Grade 3 or Grade 4 toxicity criteria will be plotted as mean values over time. Serum chemistry parameters for patients that meet Grade 3 or Grade 4 toxicity criteria from the CTCAE v4.0 for total cholesterol, low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL), and triglycerides will be summarized for each scheduled visit and overall for all post-baseline visits.

Laboratory values will be converted to the project-defined unit of measurement, as applicable, before analysis. If laboratory values are recorded as above or below a threshold (i.e. "<2", ">30",


etc.), they will be counted as missing for continuous summaries. Abnormal, clinically significant laboratory values (per Investigator judgment) will be reported and summarized as AEs.

All laboratory parameter results will be included in by-patient data listings. Reference ranges for each clinical laboratory parameter will also be summarized in a data listing.

#### 9.4 Vital Signs, Physical Findings, and Other Observations Related to Safety

## 9.4.1 Vital Signs

Baseline will be defined as the last vital sign value obtained before the first dose of study drug on Day 1; if Day 1 values are unavailable, then values obtained at the Screening Visit will be used. Observed vital sign measurements along with change from baseline for each scheduled assessment will be summarized descriptively by treatment group and visit for each vital sign variable specified in the protocol (Systolic Blood Pressure, Diastolic Blood Pressure, Pulse Rate, Respiratory Rate, and Oral Temperature). Vital signs will also be presented for each patient in a data listing.

#### 9.4.2 ECG

Observed Overall ECG Interpretations will be summarized as Normal, Abnormal and Not Clinically Significant, or Abnormal and Clinically Significant for each scheduled visit by treatment group. In addition, observed and change from baseline measurements of ECG intervals (PR, QT, QTcF, QRS, and RR) for each scheduled assessment will be summarized descriptively by treatment group and visit as well as listed within a by-patient data listing. Patients receiving study drug will be identified and summarized by treatment group and visit, as well as overall for the following clinically notable categories:

- QTcF > baseline and > 450 msec
- QTcF > baseline and > 480 msec
- QTcF > baseline and > 500 msec
- QTcF increase from baseline > 30 msec
- QTcF increase from baseline > 60 msec

## 9.4.3 Physical Examinations

A listing of physical examinations will be provided. Deteriorations from baseline on physical examination will be coded as adverse events and summarized as such.


## 10. PHARMACOKINETIC EVALUATION

# 10.1 Pharmacokinetic and Pharmacodynamic Methods

The collection status of pharmacokinetic and pharmacodynamic samples will be listed for each visit with scheduled sampling by patient using the Safety Population. Plasma concentrations of study drug may be summarized separately, as appropriate, for the Pharmacokinetic Population.


#### 11. INTERIM ANALYSES AND DATA MONITORING

When SALT data through Week 24 of treatment was available for all patients in Cohort 1 (4 mg) and Cohort 2 (8 mg), an interim analysis was performed. The purpose was to review selected efficacy and safety results in those 2 cohorts for planning purposes regarding the clinical development of the compound. While the results showed aggregate comparisons between the patients who received active CTP-543 and those who received placebo, all blinded study personnel remained blinded to treatment assignment. Since no further enrollment occurred in these 2 cohorts, there will be no adjustment for multiple treatment group comparisons. See Section 14 and 15 for summary tables and figures that were generated for this interim analysis.

A Data Monitoring Committee will monitor safety at regular intervals as defined in the DMC Charter. After the last patient in a cohort has completed the Week 12 Visit, the DMC will convene to review accumulated safety data to assess if initiation of the subsequent cohort is supported, as applicable. Specifications of data to be supplied to the Committee are outside the scope of this document. Further details are provided in the latest version of the DMC Charter.


#### 12. CHANGES TO THE ANALYSES PLANNED IN THE PROTOCOL

The following alterations were made to the original analyses planned in the protocol:

- SALT 50% reduction analysis changed from Cochran-Mantel-Haenszel Test (CMH) to  $\chi^2$  test and will not be stratified by Alopecia Areata subtype.
- VAS-S analysis method changed from CMH to ANCOVA.
- CGI-I and PGI-I analysis method changed from CMH test to  $\chi^2$  test.
- AASIS and Exploratory Question analysis method changed from ANCOVA to descriptive statistics and  $\chi^2$  test, respectively.
- Alopecia Areata subtype used as a fixed effect within the MMRM.
- TEAE definition modified so that all AEs that occur after study dosing will be counted, rather than only those that occur up to Week 24 or the Early Termination Visit.

## 13. REFERENCES

Mendoza TR, Osei JS, Shi Q, Duvic M. Development of the alopecia areata symptom impact scale. J Investig Dermatol Symp Proc. 2013 Dec;16(1):S51-2.

Olsen EA, Hordinsky MK, Price VH, et al. Alopecia areata investigational assessment guidelines--Part II. National Alopecia Areata Foundation. J Am Acad Dermatol. 2004 Sep;51(3):440-7.


## 14. LIST OF PLANNED TABLES

| Table ID | Table No. | Title | Population | Unique? | Interim<br>Analysis |
|---|---|---|---|---|---|
| DS_TAA | 14.1.1 | Summary of Patient<br>Disposition | All<br>Screened<br>Patients | Y | X |
| DS_TAB | 14.1.2 | Summary of<br>Protocol Deviations | All<br>Randomized<br>Patients | Y | |
| DM_TAA | 14.1.3 | Summary of<br>Demographics | All<br>Randomized<br>Patients | Y | X |
| DM_TAB | 14.1.4 | Summary of Baseline Characteristics | All<br>Randomized<br>Patients | Y | X |
| MH_TAA | 14.1.5 | Summary of<br>Medical History by<br>System Organ<br>Class and Preferred<br>Term | Safety<br>Population | Y | |
| EX_TAA | 14.1.6.1 | Summary of Study Drug Administration and Compliance by Treatment Group | Safety<br>Population | Y | |
| CM_TAA | 14.1.7.1 | Summary of Prior<br>Medications | Safety<br>Population | N | |
| CM_TAB | 14.1.7.2 | Summary of<br>Concomitant<br>Medications | Safety<br>Population | N | |
| EF_TAA | 14.2.1.1 | Chi-Squared<br>Analysis of<br>Responders at<br>Week 24 | Efficacy<br>Population | Y | X |
| EF_TAB | 14.2.1.2 | Chi-Squared<br>Analysis of<br>Responders at<br>Week 24 | Per Protocol<br>Population | N | |
| EF_TAC | 14.2.1.3 | Chi-Squared<br>Analysis of<br>Responders by<br>Visit | Efficacy<br>Population | N | X |
| EF_TAD | 14.2.1.4 | Chi-Squared<br>Analysis of | Per Protocol<br>Population | N | |


| | | Responders by | | | |
|---|---|---|---|---|---|
| EF_TAT | 14.2.1.5 | Visit Chi-Squared Analysis of Patients Achieving ≤10, ≤20, or ≤25 Absolute Salt Scores by Visit | Efficacy<br>Population | N | |
| EF_TAU | 14.2.1.6 | Chi-Squared Analysis of Patients Achieving ≤10, ≤20, or ≤25 Absolute Salt Scores by Visit | Per Protocol<br>Population | N | |
| EF_TAE | 14.2.1.7.1 | Summary of Total<br>SALT Scores by<br>Treatment Group<br>and Visit | Efficacy<br>Population | Y | X |
| EF_TAI | 14.2.1.7.2 | Summary of Total<br>SALT Scores of<br>Responders at<br>Week 24 by<br>Treatment Group | Efficacy<br>Population | Y | X |
| EF_TAF | 14.2.1.8 | MMRM Analysis<br>for Absolute<br>Change in SALT<br>Scores | Efficacy<br>Population | Y | X |
| EF_TAG | 14.2.1.9 | MMRM Analysis<br>for Absolute<br>Change in SALT<br>Scores | Per Protocol<br>Population | N | |
| EF_TAH | 14.2.1.10 | MMRM Analysis<br>for Relative<br>Change in SALT<br>Scores | Efficacy<br>Population | N | X |
| EF_TAS | 14.2.1.11 | MMRM Analysis<br>for Relative<br>Change in SALT<br>Scores | Per Protocol<br>Population | N | |
| EF_TAY | 14.2.1.12 | MMRM Analysis<br>for Absolute SALT<br>Scores | Efficacy<br>Population | N | |
| EF_TAZ | 14.2.1.13 | MMRM Analysis<br>for Absolute SALT<br>Scores | Per Protocol<br>Population | N | |


| | 14001 | | T CC | <u> </u> | |
|---|---|---|---|---|---|
| EF_TAJ | 14.2.2.1 | Summary of | Efficacy | | |
| | | Clinician VAS-S | Population | Y | |
| | 14222 | (mm) | E.C.C. | NT. | |
| EF_TAK | 14.2.2.2 | Summary of Patient | Efficacy | N | |
| | 11001 | VAS-S (mm) | Population | | |
| EF_TAL | 14.2.3.1 | Summary of CGI-I | Efficacy | Y | |
| | | | Population | | |
| EF_TAM | 14.2.3.2 | Summary of CGI-I | Efficacy | Y | |
| | | Improvement | Population | | |
| EF_TAN | 14.2.3.3 | Summary of CGI-I | Efficacy | N | |
| | | Worsening | Population | | |
| EF_TAO | 14.2.3.4 | Summary of PGI-I | Efficacy<br>Population | N | |
| EE TAD | 14.2.3.5 | Summary of PGI-I | Efficacy | N | |
| EF_TAP | 14.2.3.3 | Improvement | Population | 1,4 | |
| EE TAO | 14.2.3.6 | Summary of PGI-I | Efficacy | N | |
| EF_TAQ | 14.2.3.0 | Worsening | Population | 1 | |
| EF TAR | 14.2.4.1 | Summary of | Efficacy | Y | |
| Er_IAK | 14.2.4.1 | Exploratory | Population | 1 | |
| | | Questions at Week | Fopulation | | |
| | | 24 | | | |
| DD TAX | 14.2.4.2 | Shift from Baseline | Efficacy | Y | |
| EF_TAV | 14.2.4.2 | to Week 24 | Population | 1 | |
| | | Exploratory | Fopulation | | |
| | | Questions | | | |
| DD TAXY | 14.2.5.1 | Summary of | Efficacy | Y | |
| EF_TAW | 14.2.3.1 | AASIS Responses | Population | 1 | |
| DD TAX | 14.2.5.2 | Mean and Mean | Efficacy | Y | |
| EF_TAX | 14.2.3.2 | Change from | Population | 1 | |
| | | Baseline in AASIS | Population | | |
| AT TAA | 1/12 1 1 | Responses | Safety | V | v |
| AE_TAA | 14.3.1.1 | Summary of<br>Treatment- | | Y | X |
| | | | Population | | |
| | | Emergent Adverse Events | | | |
| AT TAR | 14.3.1.2 | | Safety | Y | X |
| AE_TAB | 14.5.1.2 | Summary of<br>Treatment- | Population | 1 | Λ |
| | | Emergent Adverse | Fobulation | | |
| | | Events by System | | | |
| | | Organ Class and | | | |
| | | Preferred Term | | | |
| AE TAC | 14.3.1.3 | Summary of | Safety | N | |
| AE_TAC | 14.5.1.5 | Treatment- | Population | 1 | |
| | | | Fobulation | | |
| | | Emergent Serious Adverse Events by | | | |
| | | System Organ | | | |


| | T | Class and Dusfamed | T | |
|---|---|---|---|---|
| | | Class and Preferred | | |
| | | Term | ~ 0 | |
| AE_TAD | 14.3.1.4 | Summary of All | Safety | N |
| | | Treatment- | Population | |
| | | Emergent Adverse | | |
| | | Events Leading to | | |
| | | Discontinuation of | | |
| | | Study Drug System | | |
| | | Organ Class and | | |
| | | Preferred Term | | |
| AE TAE | 14.3.1.5 | Summary of | Safety | N |
| TL_TTL | | Treatment- | Population | - |
| | | Emergent Adverse | 1 op diameter | |
| | | Events Resulting in | | |
| | | Study Dose | | |
| | | Interruption by | | |
| | | System Organ | | |
| | | Class and Preferred | | |
| | 11216 | Term | G 0 : | 3.7 |
| AE_TAF | 14.3.1.6 | Summary of | Safety | N |
| | | CTCAE Grade 3-4 | Population | |
| | | Hematology | | |
| | | Treatment- | | |
| | | Emergent Adverse | | |
| | | Events by System | | |
| | | Organ Class and | | |
| | | Preferred Term | | |
| AE TAG | 14.3.1.7 | Summary of | Safety | N |
| 1110 | | CTCAE Grade 3-4 | Population | |
| | | Serum Chemistry | <b>F</b> | |
| | | Treatment- | | |
| | | Emergent Adverse | | |
| | | Events by System | | |
| | | Organ Class and | | |
| | | Preferred Term | | |
| AD TAIL | 14.3.1.8 | | Cofoty | Y |
| AE_TAH | 14.3.1.8 | Summary of<br>Treatment- | Safety | 1 |
| | | | Population | |
| | | Emergent Adverse | | |
| | | Events by | | |
| | | Severity/Intensity, | | |
| | | System Organ | | |
| | | Class, and | | |
| | | D f 1 T | 1 | 1 |
| | | Preferred Term | | |
| AE TAI | 14.3.1.9 | Summary of | Safety | Y |
| AE_TAI | 14.3.1.9 | | Safety<br>Population | Y |


| | 1 | | T | |
|---|---|---|---|---|
| | | Events by System | | |
| | | Organ Class and<br>Preferred Term: | | |
| | | Incidence by Time<br>Interval | | |
| | 142110 | | Cafata | NT. |
| AE_TAJ | 14.3.1.10 | Summary of | Safety | N |
| | | Treatment- | Population | |
| | | Emergent Adverse | | |
| | | Events by System | | |
| | | Organ Class and | | |
| | | Preferred Term: | | |
| | | Prevalence by Time | | |
| | | Interval | | |
| AE_TAK | 14.3.1.11 | Summary of | Safety | N |
| | | CTCAE Grade 3-4 | Population | |
| | | Treatment- | | |
| | | Emergent | | |
| | | Hematology | | |
| | | Adverse Events | | |
| | | System Organ | | |
| | | Class and Preferred | | |
| | | Term: Incidence by | | |
| | | Time Interval | | |
| AE_TAL | 14.3.1.12 | Summary of | Safety | N |
| | | CTCAE Grade 3-4 | Population | |
| | | Treatment- | | |
| 1 | | | | |
| | | Emergent | | |
| | | Hematology | | |
| | | Hematology<br>Adverse Events | | |
| | | Hematology<br>Adverse Events<br>System Organ | | |
| | | Hematology<br>Adverse Events<br>System Organ<br>Class and Preferred | | |
| | | Hematology Adverse Events System Organ Class and Preferred Term: Prevalence | | |
| | | Hematology Adverse Events System Organ Class and Preferred Term: Prevalence by Time Interval | | |
| AE_TAM | 14.3.1.13 | Hematology Adverse Events System Organ Class and Preferred Term: Prevalence by Time Interval Summary of | Safety | N |
| AE_TAM | 14.3.1.13 | Hematology Adverse Events System Organ Class and Preferred Term: Prevalence by Time Interval Summary of CTCAE Grade 3-4 | Safety<br>Population | N |
| AE_TAM | 14.3.1.13 | Hematology Adverse Events System Organ Class and Preferred Term: Prevalence by Time Interval Summary of CTCAE Grade 3-4 Treatment- | • | N |
| AE_TAM | 14.3.1.13 | Hematology Adverse Events System Organ Class and Preferred Term: Prevalence by Time Interval Summary of CTCAE Grade 3-4 Treatment- Emergent Serum | • | N |
| AE_TAM | 14.3.1.13 | Hematology Adverse Events System Organ Class and Preferred Term: Prevalence by Time Interval Summary of CTCAE Grade 3-4 Treatment- Emergent Serum Chemistry Adverse | • | N |
| AE_TAM | 14.3.1.13 | Hematology Adverse Events System Organ Class and Preferred Term: Prevalence by Time Interval Summary of CTCAE Grade 3-4 Treatment- Emergent Serum Chemistry Adverse Events System | • | N |
| AE_TAM | 14.3.1.13 | Hematology Adverse Events System Organ Class and Preferred Term: Prevalence by Time Interval Summary of CTCAE Grade 3-4 Treatment- Emergent Serum Chemistry Adverse Events System Organ Class and | • | N |
| AE_TAM | 14.3.1.13 | Hematology Adverse Events System Organ Class and Preferred Term: Prevalence by Time Interval Summary of CTCAE Grade 3-4 Treatment- Emergent Serum Chemistry Adverse Events System Organ Class and Preferred Term: | • | N |
| AE_TAM | 14.3.1.13 | Hematology Adverse Events System Organ Class and Preferred Term: Prevalence by Time Interval Summary of CTCAE Grade 3-4 Treatment- Emergent Serum Chemistry Adverse Events System Organ Class and Preferred Term: Incidence by Time | • | N |
| | | Hematology Adverse Events System Organ Class and Preferred Term: Prevalence by Time Interval Summary of CTCAE Grade 3-4 Treatment- Emergent Serum Chemistry Adverse Events System Organ Class and Preferred Term: Incidence by Time Interval | Population | |
| AE_TAM AE_TAN | 14.3.1.13 | Hematology Adverse Events System Organ Class and Preferred Term: Prevalence by Time Interval Summary of CTCAE Grade 3-4 Treatment- Emergent Serum Chemistry Adverse Events System Organ Class and Preferred Term: Incidence by Time Interval Summary of | Population Safety | N |
| | | Hematology Adverse Events System Organ Class and Preferred Term: Prevalence by Time Interval Summary of CTCAE Grade 3-4 Treatment- Emergent Serum Chemistry Adverse Events System Organ Class and Preferred Term: Incidence by Time Interval | Population | |


| AE_TAO | 14.3.1.15 | Emergent Hematology Adverse Events by System Organ Class and Preferred Term: Prevalence by Time Interval Summary of Treatment- Emergent Adverse Events by Relationship to Study Drug, System Organ Class, and Preferred Term | Safety<br>Population | N | |
|---|---|---|---|---|---|
| AE_TAP | 14.3.1.16 | Summary of Treatment- Emergent Serious Adverse Events by Relationship to Study Drug, System Organ Class, and Preferred Term | Safety<br>Population | N | |
| LB_TAA | 14.3.4.1.1 | Summary of All<br>Clinical Laboratory<br>Values:<br>Hematology | Safety<br>Population | Y | X |
| LB_TAB | 14.3.4.1.2 | Summary of All<br>Clinical Laboratory<br>Values: Serum<br>Chemistry | Safety<br>Population | N | |
| LB_TAC | 14.3.4.2.1 | Summary of<br>CTCAE Grade 3-4<br>Key Clinical<br>Laboratory Values:<br>Hematology | Safety<br>Population | Y | X |
| LB_TAD | 14.3.4.2.2 | Summary of<br>CTCAE Grade 3-4<br>Key Clinical<br>Laboratory Values:<br>Serum Chemistry | Safety<br>Population | N | |
| VS_TAA | 14.3.5.1 | Vital Signs<br>Summary | Safety<br>Population | Y | |


| EG_TAA | 14.3.5.2 | 12-Lead<br>Electrocardiogram<br>Summary | Safety<br>Population | N |
|---|---|---|---|---|
| EG_TAB | 14.3.5.3 | Summary of Abnormal, Clinically Significant 12-Lead Electrocardiogram Values by Treatment Group and Visit | Safety<br>Population | Y |
| EG_TAC | 14.3.5.4 | Summary of Clinically Notable 12-Lead Electrocardiogram Values by Treatment Group and Visit | Safety<br>Population | Y |


## **15.LIST OF PLANNED FIGURES**

| Figure ID | Figure No. | Title | Population | Unique? | Interim<br>Analysis |
|---|---|---|---|---|---|
| DS_FAA | 14.1.1 | Kaplan-Meier Plot for<br>Time to Last Dose | Safety<br>Population | Y | |
| EF_FAA | 14.2.1.1 | Responders by<br>Treatment at Week 24 | Efficacy<br>Population | Y | X |
| EF_FAB | 14.2.1.2 | Responders by<br>Treatment across Time | Efficacy<br>Population | Y | X |
| EF_FAC | 14.2.1.3 | Mean SALT Scores by<br>Treatment across Time | Efficacy<br>Population | Y | X |
| EF_FAD | 14.2.1.4 | Mean Absolute Change<br>in SALT Scores by<br>Treatment across Time | Efficacy<br>Population | N | X |
| EF_FAE | 14.2.1.5 | Mean Relative Change<br>in SALT Scores by<br>Treatment across Time | Efficacy<br>Population | N | X |
| LB_FAA | 14.3.4.1.1 | Key Clinical Laboratory<br>Values: Hematology<br>Parameters | Safety<br>Population | Y | |


## **16. LIST OF PLANNED DATA LISTINGS**

| Listing ID | Listing<br>No. | Title | Population | Unique? | Interim<br>Analysis |
|---|---|---|---|---|---|
| RN LAA | 16.1.1 | Randomization | All Randomized | Y | |
| _ | | Codes | Patients | | |
| LB_LAA | 16.1.10.1 | Clinical Laboratory<br>Reference Range | N/A | Y | |
| DS_LAA | 16.2.1.1 | Patient Disposition | All Randomized<br>Patients | Y | |
| DS_LAB | 16.2.1.2 | Screen Failures | | Y | |
| DS_LAC | 16.2.1.3 | Screen Failures Prior to Amendment 2 | | N | |
| DS_LAD | 16.2.1.4 | Patient Visits | All Randomized<br>Patients | Y | |
| DS_LAE | 16.2.2 | Protocol Deviations | All Randomized<br>Patients | Y | |
| DS_LAF | 16.2.3 | Analysis Sets | All Randomized<br>Patients | Y | |
| DM_LAA | 16.2.4.1 | Patient Demographic and Baseline Characteristics | All Randomized<br>Patients | Y | |
| DM_LAB | 16.2.4.2 | Alopecia Areata<br>History | All Randomized<br>Patients | Y | |
| MH_LAA | 16.2.4.3 | Medical History | Safety Population | Y | |
| CM_LAA | 16.2.4.4 | Prior and<br>Concomitant<br>Medications | Safety Population | Y | |
| EX_LAA | 16.2.5.1 | Treatment<br>Compliance | Safety Population | Y | |
| EX_LAB | 16.2.5.2 | Dosing Exceptions | Safety Population | Y | |
| EF_LAA | 16.2.6.1 | SALT Score | Efficacy<br>Population | Y | |
| EF_LAB | 16.2.6.2 | SALT Photographs | Efficacy<br>Population | Y | |
| EF_LAC | 16.2.6.3 | Clinician and<br>Patient VAS-S | Efficacy<br>Population | Y | |
| EF_LAD | 16.2.6.4 | CGI-I and PGI-I | Efficacy<br>Population | Y | |
| EF_LAE | 16.2.6.5 | AASIS | Efficacy<br>Population | Y | |


| EF_LAF | 16.2.6.6 | Exploratory | Efficacy | N |
|---|---|---|---|---|
| | | Questions | Population | |
| AE_LAA | 16.2.7.1 | All Adverse Events | Safety Population | Y |
| AE_LAB | 16.2.7.2 | Serious Adverse<br>Events | Safety Population | N |
| AE_LAC | 16.2.7.3 | Adverse Events<br>Related to Study<br>Drug | Safety Population | N |
| AE_LAD | 16.2.7.4 | Adverse Events Leading to Study Drug Discontinuation | Safety Population | N |
| AE_LAE | 16.2.7.5 | Adverse Events Leading to Study Drug Interruption | Safety Population | N |
| AE_LAF | 16.2.7.6 | Adverse Events<br>Leading to Death | Safety Population | N |
| AE_LAG | 16.2.7.7 | Pregnancy | Safety Population | N |
| PE_LAA | 16.2.8 | Physical<br>Examinations | Safety Population | Y |
| LB_LAB | 16.2.9.1 | Clinical Laboratory<br>Data: Hematology | Safety Population | Y |
| LB_LAC | 16.2.9.2 | Clinical Laboratory<br>Data: Serum<br>Chemistry | Safety Population | N |
| VS_LAA | 16.2.10.1 | Vital Signs | Safety Population | Y |
| EG_LAA | 16.2.10.2 | 12-Lead<br>Electrocardiogram | Safety Population | Y |
| PK_LAA | 16.2.10.3 | Pharmacokinetic<br>Blood Samples | Pharmacokinetic<br>Population | Y |
| PD_LAA | 16.2.10.4 | Pharmacodynamic<br>Blood Samples | Pharmacokinetic<br>Population | Y |


## 17. APPENDICES

# 17.1 Study Flow Chart




## 17.2 Schedule of Events

| | Screening | Randomization | Treatment Period | | | | Safety<br>Follow-Up | |
|---|---|---|---|---|---|---|---|---|
| | Day -28 to Day -112 | Day 1 <sup>1</sup> | Week 2, 6 | Week 4, 8 | Week 12 | Week 16, 20 | Week 24 <sup>11</sup> | Week 28 |
| Event | (Visit 1) | (Visit 2) | (Visit 3, 5) | (Visit 4, 6) | (Visit 7) | (Visit 8, 9) | (Visit 10) | (Visit 11) <sup>13</sup> |
| Informed consent | X | | | | | | | |
| Eligibility assessment | X | X | | | | | | |
| Demographics | X | | | | | | | |
| Medical history | X | X | | | | | | |
| Randomization | | X | | | | | | |
| Physical examination | X | X | | | | | X | X |
| Brief physical examination | | | | X | X | X | | |
| Height | X | | | | | | | |
| Weight | X | X | | X | X | X | X | X |
| Pregnancy test <sup>2</sup> | X | X | | X | X | X | X | |
| Tuberculosis test | X | | | | | | | |
| Clinical laboratory testing <sup>3,8</sup> | $X^4$ | X | X | X | X | X | X | X |
| Lipid assessment <sup>5</sup> | | X | | | X | | X | X |
| HBV and HCV test | X | | | | | | | |
| Pharmacokinetic blood sampling | | $X^6$ | $X^6$ | $X^6$ | | | $X^6$ | |
| Pharmacodynamic blood sampling | | $X^7$ | $X^7$ | $X^7$ | | | $X^7$ | |
| 12-lead electrocardiogram | X | X | | X | X | X | X | X |
| Vital signs | X | X | | X | X | X | X | X |
| Severity of Alopecia Tool assessment <sup>9</sup> | X | X | | X | X | X | X | |
| Photographs | X | X | | X | X | X | X | |
| Clinician Visual Analog Scale – Severity <sup>9</sup> | | X | | | X | | X | |
| Clinician Global Impression of Improvement9 | | | | | X | | X | |
| Patient Visual Analog Scale - Severity | | X | | | X | | X | |
| Patient Global Impression of Improvement | | | | | X | | X | |
| AASIS and exploratory questions | | X | | | | | X | |
| Dispense study drug | | X | | X | X | X | | |
| Study drug accountability | | | | X | X | X | X | |
| Adverse events <sup>10</sup> | X | X | X | X | X | X | X | X |
| Concomitant medications <sup>10</sup> | X | X | X | X | X | X | X | X |

Version: 2.0 Page **48** of **50** 

#### CONFIDENTIAL

### Statistical Analysis Plan 07 May 2019

| AASIS = Alopecia Areata Symptom Impact Scale; HBV= hepatitis B virus; HCV = hepatitis C virus | Ī |
|---|---|
| All subsequent visits and week increments should be based on the date of Visit 2. All | ı |
| visit windows are ±3 days. | 9 |

- <sup>2</sup> Serum pregnancy test only for females of childbearing potential.
- <sup>3</sup> Includes hematology and serum chemistry.
- <sup>4</sup> Will include thyroid stimulating hormone and hemoglobin A1c at Screening only.
- <sup>5</sup> Includes total cholesterol, low-density lipoprotein, high-density lipoprotein, and triglycerides.
- <sup>6</sup> Collected at Day 1 and Week 4 (pre-dose, and post-dose at end of visit), and Weeks 2 (pre-dose with clinical labs), and Weeks 8, 24 (post-dose at end of visit).
- Collected at Day 1 and Week 2 (pre-dose with clinical labs), and Weeks 4, 8, 24 (post-dose at end of visit).<sup>8</sup> Collected pre-dose.
- <sup>9</sup> Should be performed by the same rater for the patient for the duration of the study.
- <sup>10</sup> Collection is ongoing.
- <sup>11</sup> Also serves as the Early Termination Visit for patient withdrawal.
- Randomization/Day 1 may occur any time after Screening laboratory results are available and reviewed by the Investigator.
- The Safety Follow-Up Visit is intended for those patients in Cohort 1 and Cohort 2, and those patients in Cohort 3 who do not roll over into the Open-label Extension.


## 18. ATTACHMENTS

Attachment A: "CP543.2001 - TLF Shells" - Shells for Planned Tables, Figures, and Listings
